CLINICAL TRIAL: NCT02515890
Title: Modulation of Long-term Memory by the Experience of Pain During Sedation With Anesthetics
Brief Title: Memory Modulation by Pain During Anesthesia
Acronym: MMA
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Pittsburgh (Other)
Collaborators: Foundation for Anesthesia Education and Research (Other)
Responsible Party: Principal Investigator, Keith M. Vogt, MD, PhD, Assistant Professor, University of Pittsburgh
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: PRO14050609
Record Dates: First submitted 2015-08-03; First posted 2015-08-05 (Estimated); Results first posted 2020-07-01 (Actual); Last update posted 2020-07-01 (Actual); Status verified 2020-06

CONDITIONS: Amnesia; Pain; Anesthesia
Keywords: midazolam; dexmedetomidine; memory; ketamine
MeSH Terms: conditions — Amnesia; Pain | interventions — Dexmedetomidine; Midazolam; Transcutaneous Electric Nerve Stimulation; Ketamine

STUDY DESIGN:
Intervention Model Description: There are 3 single drug arms completed by a few participants. The majority of participants participated in a crossover design with two drugs, midazolam & ketamine.
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: Yes

ARMS (5):
- Dexmedetomidine Only (Experimental): All subjects receive saline (control), followed by a dexmedetomidine infusion. They also experience intermittent experimental pain delivered by peripheral nerve stimulation.
  Interventions: Drug: Dexmedetomidine; Device: Peripheral nerve stimulation
- Midazolam Only (Experimental): Subjects receive saline (control), followed by midazolam infusion. They also experience intermittent experimental pain delivered by peripheral nerve stimulation.
  Interventions: Drug: Midazolam; Device: Peripheral nerve stimulation
- Ketamine Only (Experimental): All subjects receive saline (control), followed by ketamine infusion. They also experience intermittent experimental pain delivered by peripheral nerve stimulation.
  Interventions: Device: Peripheral nerve stimulation; Drug: Ketamine
- Saline/Midazolam/Saline/Ketamine (Experimental): All subjects receive saline (control), followed by midazolam infusion. They also experience intermittent experimental pain delivered by peripheral nerve stimulation.
  Subjects then returned at least 1 week later for another set of experimental sessions with the same design, however the saline was followed by ketamine infusion.
  Interventions: Drug: Midazolam; Device: Peripheral nerve stimulation; Drug: Ketamine
- Saline/Ketamine/Saline/Midazolam (Experimental): All subjects receive saline (control), followed by ketamine infusion. They also experience intermittent experimental pain delivered by peripheral nerve stimulation.
  Subjects then returned at least 1 week later for another set of experimental sessions with the same design, however the saline was followed by midazolam infusion.
  Interventions: Drug: Midazolam; Device: Peripheral nerve stimulation; Drug: Ketamine

INTERVENTIONS:
Drug: Dexmedetomidine — Selected subjects received this drug during a portion of the study
  Other Names: Precedex
  Arms: Dexmedetomidine Only
Drug: Midazolam — Selected subjects received this drug during a portion of the study
  Other Names: Versed
  Arms: Midazolam Only; Saline/Ketamine/Saline/Midazolam; Saline/Midazolam/Saline/Ketamine
Device: Peripheral nerve stimulation — Experimental acute pain stimulus was delivered using a nerve stimulator. These painful shocks were paired randomly with some of the auditory experimental cues.
  Other Names: electric nerve stimulation
Drug: Ketamine — Selected subjects received this drug during a portion of the study
  Other Names: Ketalar
  Arms: Ketamine Only; Saline/Ketamine/Saline/Midazolam; Saline/Midazolam/Saline/Ketamine

SUMMARY:
The purpose of this study is to determine the effects of pain on facilitating long-term auditory memory in the presence and absence of distinct intravenous anesthetics. The ability to identify previously presented words from a list assessed the degree of memory formation. In a subset of subjects, functional magnetic resonance imaging was used to identify the neural correlates of memory inhibition or facilitation by the combination of pain and anesthetic used.

DETAILED DESCRIPTION:
This study adds specific details to the current incomplete body of knowledge examining the effect of pain on memory formation under the influence of anesthetic agents.

Pain and anesthetic agents were administered as experimental variables in this study. Healthy adult subjects were played repeated lists of words and performed several decision-making tasks that encourage memory encoding. Some words were consistently paired with painful electric shock, and was anticipated to improve subsequent memory performance specifically for those items. The same experiment was repeated in all subjects during the administration of 1-2 possible agents that reduce memory formation: dexmedetomidine, a predominantly sedative agent, and midazolam, a well-known amnestic agent, and ketamine, a well-known dissociative analgo-sedative. The extent to which pain modulates memory performance under the effects of the anesthetic agents was the primary outcome of interest.

Further, a subset of the subjects performed the same experimental procedures while undergoing functional magnetic resonance imaging, which continuously reflects neuronal activity throughout the brain. Classic memory areas were predicted to be activated by the auditory processing task, but how these neural circuits change under the two anesthetic agents with the concomitant experience of pain were of interest. It was anticipated that pain recruits a parallel memory pathway using limbic structures, known for their involvement in fear conditioning. Additionally, stronger and more diffuse cortical processing likely occurs with concomitant pain, as level of sedation was reduced by this strong stimulus. Discovering the anatomic correlates specific to each experimental variable (pain and anesthetic), and their interplay, may help refine our model of brain function during the dynamics of pain and sedation.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adult volunteers, with normal memory and hearing, whose native language is English

Exclusion Criteria:

* pregnancy
* significant memory or hearing loss
* sleep apnea
* chronic pain
* metal or electronic implants
* claustrophobia
* Currently taking: antidepressants, anti-psychotics, antihistamines, anti-anxiety medication, stimulants, sleep-aids, or pain medication

Ages: 18 Years to 39 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 32 (Actual)
Dates: Start 2015-11-19 (Actual); Primary Completion 2018-12-12 (Actual); Study Completion 2018-12-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Keith M Vogt, MD, PhD, Principal Investigator — University of Pittsburgh
Locations (1):
- University of Pittsburgh, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Yes
Data will be published. After all analysis and dissemination is complete, functional images will be shared via data repository.

RESULTS

PARTICIPANT FLOW:
Groups:
- Dexmedetomidine: subjects received dexmedetomidine and saline (control)
- Midazolam: subjects received midazolam and saline (control)
- Ketamine: subjects received ketamine and saline (control)
- Drug Order A: Subjects received saline (control) and midazolam during their first set of experimental sessions, and then received saline (control) and ketamine during a second set of sessions
- Drug Order B: Subjects received saline (control) and ketamine during their first set of experimental sessions, and then received saline (control) and midazolam during a second set of sessions
Period: Overall Study
Arm/Group | Dexmedetomidine | Midazolam | Ketamine | Drug Order A | Drug Order B
Started | 7 | 4 | 5 | 8 | 8
Completed | 7 | 4 | 5 | 8 | 8
Not Completed | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Dexmedetomidine Only: All subjects received saline (control) followed by dexmedetomidine infusion while performing memory task and receiving intermittent painful electric nerve stimulation.
- Midazolam Only: All subjects received saline (control) followed by midazolam infusion while performing memory task and receiving intermittent painful electric nerve stimulation.
- Ketamine Only: All subjects received saline (control) followed by ketamine infusion while performing memory task and receiving intermittent painful electric nerve stimulation.
- Drug Order A: All subjects received saline (control) followed by midazolam infusion while performing memory task and receiving intermittent painful electric nerve stimulation on their first experimental visit.
  For another experimental session, all subjects received saline (control) followed by ketamine infusion while performing memory task and receiving intermittent painful electric nerve stimulation.
- Drug Order B: All subjects received saline (control) followed by ketamine infusion while performing memory task and receiving intermittent painful electric nerve stimulation on their first experimental visit.
  For another experimental session, all subjects received saline (control) followed by midazolam infusion while performing memory task and receiving intermittent painful electric nerve stimulation.
- Total: Total of all reporting groups
Arm/Group | Dexmedetomidine Only | Midazolam Only | Ketamine Only | Drug Order A | Drug Order B | Total
Number analyzed (Participants) | 7 | 4 | 5 | 8 | 8 | 32
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 7 | 4 | 5 | 8 | 8 | 32
  >=65 years | 0 | 0 | 0 | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 2 | 1 | 3 | 5 | 14
  Male | 4 | 2 | 4 | 5 | 3 | 18
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 7 | 4 | 5 | 8 | 8 | 32

OUTCOME MEASURES:

1. Primary Outcome: Memory Testing
Description: Subjects completed the Remember, Know, New (RKN) task during next day testing. Their d' memory score was calculated based on their ability to discriminate between previously heard words and new words. A higher d' score indicates stronger recollection. D' scores were compared across the control condition (saline) and the drug conditions dexmedetomidine, midazolam, and ketamine. Performance was also calculated according to words associated with Pain and No Pain conditions.
Time Frame: At memory testing 1 day later
Population: The overall number analyzed for each drug condition represents the number of observations for that drug, which doesn't directly correspond to study arms. All participants received a saline control condition with their drug condition. Therefore, there were 48 saline observations (saline d' scores) which includes observations from all 5 study arms.
Measure: Mean (Standard Error); unit: d' score
Units Other Than Participants: number of observations for each drug
Groups:
- Dexmedetomidine: Subjects assigned to receive dexmedetomidine as part of the study
- Midazolam: Subjects assigned to receive midazolam as part of the study. Includes subjects from groups Midazolam Only, Drug Order A, and Drug Order B
- Ketamine: Subjects assigned to receive ketamine as part of the study. Includes subjects from groups Ketamine Only, Drug Order A, and Drug Order B
- Saline: All subjects subjects received saline as a control condition during their study visits. Includes subjects from Dexmedetomidine Only, Midazolam Only, Ketamine Only, Drug Order A, and Drug Order B.
Arm/Group | Dexmedetomidine | Midazolam | Ketamine | Saline
Number analyzed (Participants) | 7 | 4 | 5 | 16
Number analyzed (number of observations for each drug) | 7 | 20 | 21 | 48
d' score
  All Conditions | 1.20 (.27) | .56 (.05) | .82 (.07) | 1.18 (.07)
  No Pain Condition | 1.12 (.35) | .55 (.06) | .85 (.11) | 1.18 (.10)
  Pain Condition | 1.28 (.43) | .57 (.06) | .78 (.10) | 1.10 (.10)

ADVERSE EVENTS:
Time Frame: up to 18 days after the final experimental session
Groups:
- Dexmedetomidine Only: Dexmedetomidine: Subjects received this drug during a portion of the study
- Midazolam Only: Midazolam: Subjects received this drug during a portion of the study
- Ketamine Only: Ketamine: Subjects received this drug during a portion of the study
  All adverse events for Ketamine Only subjects were experienced during ketamine administration.
- Drug Order A: Midazolam: Subjects received this drug during a portion of the study
  Ketamine: Subjects received this drug during a portion of the study
  These drugs were given on separate visits, occurring at least 14 days apart.
  All adverse events for Drug Order A subjects were experienced during ketamine administration.
- Drug Order B: Ketamine: Subjects received this drug during a portion of the study
  Midazolam: Subjects received this drug during a portion of the study
  These drugs were given on separate visits, occurring at least 14 days apart.
  All adverse events for Drug Order B subjects were experienced during ketamine administration.
Arm/Group | Dexmedetomidine Only | Midazolam Only | Ketamine Only | Drug Order A | Drug Order B
All-Cause Mortality (participants affected / at risk) | 0/7 | 0/4 | 0/5 | 0/8 | 0/8
Serious Adverse Events (participants affected / at risk) | 0/7 | 0/4 | 0/5 | 0/8 | 0/8
Other Adverse Events (participants affected / at risk) | 0/7 | 0/4 | 1/5 | 1/8 | 1/8
OTHER ADVERSE EVENTS (reported when occurring in more than 3.70% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Dexmedetomidine Only (N=7) | Midazolam Only (N=4) | Ketamine Only (N=5) | Drug Order A (N=8) | Drug Order B (N=8)
Nausea and vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) — Participants who experienced adverse events (both those in the Ketamine Only group and in Drug Order A) reported the adverse event during ketamine administration.
Dysphoria (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) — The participant from Drug Order B experienced the adverse event during the ketamine administration

LIMITATIONS AND CAVEATS:
Functional imaging results are being prepared for publication.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (3):
  • Statistical Analysis Plan (2020-04-24): https://cdn.clinicaltrials.gov/large-docs/90/NCT02515890/SAP_000.pdf
  • Informed Consent Form (2018-02-23): https://cdn.clinicaltrials.gov/large-docs/90/NCT02515890/ICF_001.pdf
  • Study Protocol (2019-01-30): https://cdn.clinicaltrials.gov/large-docs/90/NCT02515890/Prot_002.pdf